CLINICAL TRIAL: NCT06483984
Title: Physiological Effects of Novel Noninvasive Ventilation Facemasks Favoring Carbon Dioxide Washout in Patients With Hypercapnic Respiratory Failure
Brief Title: Noninvasive Ventilation Facemasks Favoring Carbon Dioxide Washout
Acronym: MASHUP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6462
Record Dates: First submitted 2024-06-17; First posted 2024-07-03 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation; Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facemask 'Nivairo' (Active Comparator): Oronasal mask for noninvasive ventilation
  Interventions: Device: Noninvasive ventilation
- Bridge-free facemask 'Visairo' (Experimental): Bridge-free facemask for noninvasive ventilation. This Bridge-Free NIV contacts the patient's nose only on the nostrils
  Interventions: Device: Noninvasive ventilation
- Facemask 'Optiniv' (Experimental): Facemask for noninvasive ventilation favoring carbon dioxide washout
  Interventions: Device: Noninvasive ventilation

INTERVENTIONS:
Device: Noninvasive ventilation — Respiratory support with a facemask connected to a ventilator through a heated humidifier. Ventilator will be set in the pressure support mode.
  Other Names: Positive-pressure ventilation

SUMMARY:
The objective of this randomized cross-over trial is to assess the physiological effects of three different facemasks for noninvasive ventilation (Nivairo, Visairo, Optiniv) in patients with acute hypercapnic respiratory failure

ELIGIBILITY:
Inclusion Criteria:

Acute respiratory failure with

* PaCO2 ≥ 45 mmHg;
* Arterial pH < 7.35;
* Signed written informed consent

Exclusion Criteria:

* Respiratory rate < 12 bpm;
* Immediate need for intubation;
* Haemodynamic instability (Systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg) and/or lactic acidosis (lactate >5 mmol/L) and/or clinically diagnosed shock;
* Metabolic Acidosis;
* Recent head surgery or anatomy that prevent the application of facemasks;
* Any contraindications to oesophageal balloon insertion and/or electrical impedance tomography (EIT) belt placement.
* Any contraindications to facemask noninvasive ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic work of breathing | 45 minutes
  Simplified pressure-time-product per minute of the transdiaphragmatic pressure

SECONDARY OUTCOMES:
Normalized metabolic work of breathing | 45 minutes
  Simplified pressure-time-product per minute of the transdiaphragmatic pressure normalized to arterial carbon dioxide divided by 45 mmHg
Inspiratory effort, expressed in cmH2O | 45 minutes
  Positive inspiratory deflection of transdiaphragmatic pressure
Corrected minute ventilation | 45 minutes
  Minute ventilation assessed with electrical impedence tomography, normalized to normalized to arterial carbon dioxide divided by 45 mmHg
Dyspnea | 45 minutes
  Dyspnoea, defined according to visual analog scale of dyspnea (0-10, where 10 represents worst perceivable dyspnea).
Discomfort | 45 minutes
  Discomfort, defined according to visual analog scale of discomfort (0-10, where 10 represents worst perceivable discomfort).
End-expiratory lung volume | 45 minutes
  Global impedance-derived end-expiratory lung volume (EELI), measured with electrical impedance tomography
Regional End-expiratory lung volume | 45 minutes
  Regional (ventral-midventral-middorsal-dorsal) impedance-derived end-expiratory lung volume (EELI), measured with electrical impedance tomography
Arterial carbon dioxide, expressed in mmHg | 45 minutes
  Arterial carbon dioxide, measured with arterial blood gas analysis
Arterial acid-base state | 45 minutes
  Arterial pH, measured with arterial blood gas analysis
Recuitment of expiratory muscles, expressed in cmH2O of gastric pressure | 45 minutes
  Expiratory increases in gastrinc pressure
Tidal volume distribution | 45 minutes
  Tidal volume distribution in the different lung regions (ventral-midventral-middorsal-dorsal),assessed with electrical impedance tomography

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Antonelli, MD, Study Chair — Catholic University of the Sacred Heart
Locations (2):
- Italy (2):
  - General intensive care unit, Fondazione Policlinico A. Gemelli IRCCS, Roma
  - Fondazione Policlinico Universitaro A. Gemelli IRCCS, Rome